CLINICAL TRIAL: NCT01974609
Title: A Randomized, Controlled Trial Comparing Combination Therapy of Ibuprofen + Acetaminophen Versus Hydrocodone + Acetaminophen for the Treatment of Pain After Carpal Tunnel Surgery
Brief Title: Narcotic vs. Non-narcotic Pain Study Protocol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Horizon Health Network (Other)
Collaborators: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other); University of Michigan (Other); Jefferson Medical College of Thomas Jefferson University (Other); McGill University (Other); University of Western Ontario, Canada (Other); Sanford Health (Other); Carilion Clinic (Other)
Responsible Party: Principal Investigator, Don Lalonde MD, MD, Horizon Health Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Narcotic vs. Non-narcotic Pain
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Carpal Tunnel
Keywords: pain relief; narcotic pain relief; non-narcotic pain relief; post-operative pain relief; carpal tunnel
MeSH Terms: conditions — Median Neuropathy | interventions — Narcotics; oxycodone-acetaminophen; Analgesics, Non-Narcotic; Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Narcotic (Experimental): Hydrocodone + acetaminophen 4 times per day 1 week after surgery
  Interventions: Drug: Narcotic
- non-narcotic (Active Comparator): ibuprofen + acetaminophen 4 times per day 1 week after surgery
  Interventions: Drug: non-narcotic

INTERVENTIONS:
Drug: Narcotic — Hydrocodone 5mg + acetaminophen 325 mg
  Other Names: Hydrocodone/acetaminophen
  Arms: Narcotic
Drug: non-narcotic — ibuprofen 600mg + acetaminophen 325 mg
  Other Names: ibuprofen + acetaminophen
  Arms: non-narcotic

SUMMARY:
The purposes of this noninferiority randomized clinical trial are to:

1. determine whether the most commonly used commonly used non-narcotic analgesic (ibuprofen 600 mg + acetaminophen 325 mg) provides pain relief that is not unacceptably worse than the most commonly prescribed narcotic containing analgesic (hydrocodone 5 mg. + acetaminophen 325 mg, equivalent to Norco 5/325) in patients undergoing carpal tunnel release.
2. Determine whether the following covariates affect pain level following surgery or medication usage: gender, country (US/Canada), pre-operative CTS symptoms, site, workers compensation status and employment status (employed/self-employed/unemployed-able to work/unemployed-unable to work)

DETAILED DESCRIPTION:
Participants will be provided with forms by site coordinators and will be provided in person instruction on how to fill out the pain intensity scores, the pain interference scores, the pain medication diary, and the final pain relief assessment form.

Medications will be identified only by number and will be available to the participant after standard instruction on use of medications is provided by the surgeon or research associate. Patients will be instructed - verbally and written - to take the study medication (2 capsules per dose) up to four times per day as needed for pain for 1 week or until pain free.

If patients experience intolerable discomfort, they will be able to contact personnel (24 hours on call) associated with the study to receive an alternate analgesic. The surgeon will determine if the patient is taking the maximum dose and then prescribe additional study drug or a non-study drug as an alternative. If the patient receives pain medication outside of the study protocol, the medication will be recorded, this will be recorded as a protocol violation. If this occurs in more than 20 people during the trial a per-protocol and efficacy analysis will be considered.

Participants will return to see the surgeon or designate between post-operative day 7 and 14 to return their diary, unused medication, and post-operative pain satisfaction survey. Participants will be specifically asked about: any adverse events, compliance with the program and the reason for any deviation and any other analgesic medication taken during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective a primary carpal tunnel release will be considered eligible

Exclusion Criteria:

* Patients wil be excluded for any of the following:
* previously enrolled in this study (for carpal tunnel surgery on the other hand);
* history of chronic opioid use;
* documented or suspected substance abuse;
* individuals currently on daily use of ibuprofen, acetaminophen or other pain altering medication including medications like Neurontin (gabapentin) and Ultram (tramadol)
* individuals with documented or suspected chronic pain syndrome;
* reported allergy or adverse reaction to hydrocodone, acetaminophen, or ibuprofen;
* those with a history or symptoms of any significant medical problem in the last year (i.e., arrhythmia, impaired cardiovascular function, gastrointestinal bleeding, liver disease, renal disease);
* patients with active peptic ulcer disease (history of severe heartburn);
* symptoms of infection with initial enrollment;
* pregnant or lactating women;
* those with a diagnosis of cognitive impairment;
* patients unable or unwilling to provide informed consent for surgery or enrollment in a clinical trial;
* patients unable or unwilling to fill out the forms or understand the consent form
* prior carpal tunnel surgery on the hand to be operated on
* individuals currently taking Coumadin, Plavix, or medications that increase bleeding; or
* patients with other medical or psychological health conditions that preclude then from receiving either intervention or returning for follow-up visits

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2016-03; Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Pain relief | 7-15 days
  1. Determine whether the most commonly used nonnarcotic analgesics (ibuprofen 600 mg + acetaminophen 325 mg) provide pain relief that is not unacceptably worse than the most commonly prescribed narcotic containing analgesic (hydrocodone 5 mg + acetaminophen 325 mg, equivalent to Norco® 5/325) in patients undergoing carpal tunnel release.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Lalonde, MD, Principal Investigator — Saint John, NB
Locations (7):
- United States (3):
  - The Philadelphia Hand Center, Philadelphia, Pennsylvania
  - Sanford orthopedics and Sports Medicine-Sioux Falls, Sioux Falls, South Dakota
  - CarilionClinic, Roanoke, Virginia
- Canada (4):
  - Horizon Health Network, Saint John, New Brunswick
  - Lawson Health Research Institute, London, Ontario
  - University of Western Ontario, Canada, London, Ontario
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lalonde DH, Lalonde JF, MacDermid JC, Chung KC, Gan BS, Mierisch C, Van Demark RE Jr, Luc M. Time to Stop Routinely Prescribing Opiates after Carpal Tunnel Release. Plast Reconstr Surg. 2022 Mar 1;149(3):651-660. doi: 10.1097/PRS.0000000000008834. PMID 35041636